CLINICAL TRIAL: NCT01183117
Title: A Clinical Investigation of SM-01 Stenting Versus PTA for the Treatment of Superficial Femoral Artery Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson K.K. Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SM-01
Record Dates: First submitted 2010-08-01; First posted 2010-08-17 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Peripheral Vascular Diseases
MeSH Terms: conditions — Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SM-01 (Experimental)
  Interventions: Device: SM-01
- PTA (Active Comparator)
  Interventions: Device: PTA

INTERVENTIONS:
Device: SM-01 — SM-01 is a self-expandable, crush recoverable stent with a diameter larger than that of the arterial lumen. The stent is indicated for use in a vessel with a diameter 1 to 2 mm smaller than the nominal stent diameter. This stent will open to the diameter of the artery and will continue to apply expanding force on the artery.
  Arms: SM-01
Device: PTA — balloon angioplasty
  Arms: PTA

SUMMARY:
The main objective is to evaluate the safety and efficacy of SM-01 stenting (Cordis S.M.A.R.T.™ Nitinol Stent System) for the treatment of SFA lesions as compared to PTA (balloon angioplasty). If SM-01 is used in a PTA-bailout patient, the case will be assessed separately.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 20 years.
2. Symptomatic leg ischemia by Rutherford Classification (category1, 2, or 3).
3. Lesion length >= 40 mm to <= 150 mm. (must be treatable with no more than two SM-01 stents. Overlap should be about 1cm if two stents are used)
4. Reference vessel diameter (RVD) >= 4.0 mm and <= 7.0 mm.
5. All lesions are to be located >= 3.0 cm proximal to the superior edge of the patella, and >= 1.0 cm distal to the SFA / PFA bifurcation.
6. >= 50% stenosis or total occlusion.
7. Patent infrapopliteal and popliteal arteries, i.e., single-vessel runoff or better with at least one of three vessels patent (< 50% stenosis) to the ankle or foot.
8. Patient or legally authorized representative must provide written informed consent prior to initiation of study procedures.
9. A patient with bilateral obstructive SFA disease is eligible for enrollment into the study. If a patient with bilateral disease is enrolled, the target limb will be the more severe limb. The more severe limb will be selected according to clinical symptomatology. If clinical symptomatology is similar, the more clinically severe lesion will be selected. The contralateral procedure should not be done until at least 30 days after the index procedure of the more severe limb was attempted.

Exclusion Criteria:

1. Recent hemorrhagic disease within the past 3 months.
2. Aneurysm in the SFA or popliteal artery.
3. Acute limb occlusion.
4. Procedures which are pre-determined to require stent-in-stent placement to obtain patency, such as severe calcification which is resistant to stenting, or for in-stent restenosis.
5. Poor iliac or common femoral "inflow".(However, intervention to restore adequate blood flow prior to the treatment of the study lesion is allowed.)
6. Known allergies to aspirin, heparin, or ticlopidine, or bleeding diathesis.
7. Patients unable or unwilling to tolerate anticoagulant or antiplatelet therapy.
8. Patients unable or unwilling to tolerate contrast agents used in intravascular procedures.
9. Allergic to nitinol or tantalum.
10. Women who are pregnant or lactating, or of child bearing potential, or with a desire to be a parent during the study period.
11. Significant vessel tortuosity or other parameters prohibiting access to the lesion or which would prevent delivery of the stent device.
12. Revascularization involving the same limb 30 days prior to the index procedure or a planned re-vascularization within 30 days after the index procedure.
13. Previously implanted stent(s) at the same site in the artery to be treated.
14. Requiring stent placement in the distal SFA or popliteal artery.
15. Presence of a femoral artificial graft.
16. History of participating in any other clinical study within 1 year.
17. Life expectancy less than 3 years, or any other factors preventing clinical follow-up.
18. Receiving dialysis or immunosuppressant therapy
19. Serum creatinine level >= 2.0 mg/dL before procedure.
20. A principal investigator or a co-principal investigator determines that patient is unsuitable for this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Non-TVF(Target-vessel failure) rate | 12 Months
  The primary endpoint will be freedom from TVF defined as any events of clinical driven (confirmed by duplex ultrasound or angiography) TLR/TVR, procedure failure, amputation of the target lesion's leg, procedure or device related death, occlusion of target lesion, or > 70% restenosis of target lesion.

SECONDARY OUTCOMES:
Procedure Success rate | 12 Months
Procedure Success rate for Bailout | 12 Months
Difference between pre and post proceduer of ABI | 12 Months
Difference between pre and post procedure of Rutherford Categories | 12 Months
Non-TLR/TVR rate | 12 Months
Primary Patency rate | 12 Months
Stent Fracture rate | 12 Months
Difference between pre and post procedure of QOL (SF-36) | 12 Months
Major Clinical Event rate | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Hidehiko Hara, MD, Principal Investigator — Toho University Ohashi Medical Center
Locations (1):
- Toho University Ohashi Medical Center, Meguro-ku, Tokyo, Japan

REFERENCES:
- [Derived] Iida O, Urasawa K, Komura Y, Soga Y, Inoue N, Hara H, Yajima J, Nakamura S, Ohki T, Ando H, Hirano K, Horita Y, Kichikawa K, Yokoi Y, Miyamoto A, Nakamura M, Takahara M, Mano T, Nanto S. Self-Expanding Nitinol Stent vs Percutaneous Transluminal Angioplasty in the Treatment of Femoropopliteal Lesions: 3-Year Data From the SM-01 Trial. J Endovasc Ther. 2019 Apr;26(2):158-167. doi: 10.1177/1526602819826591. Epub 2019 Jan 31. PMID 30702021